CLINICAL TRIAL: NCT05281003
Title: A Pilot Study of Hypoxia as a Potential Resistance Mechanism to PD-1 Checkpoint Blockade Therapy in Neoadjuvant Treatment of Esophageal Squamous Cell Carcinoma (HYPERION)
Brief Title: Pembrolizumab Plus Chemo in Neoadjuvant Treatment of Esophageal Squamous Cell Carcinoma (Eastern Cooperative Thoracic Oncology Projects 2004, ECTOP-2004)
Acronym: HYPERION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Haiquan Chen, Chief, Department of Thoracic Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTSP60942
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death Receptor Ligand 1 (PDL1, PD-L1); Esophageal Neoplasms; Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Pembrolizumab; Antineoplastic Agents; Antineoplastic Agents, Immunological; Immune Checkpoint Inhibitors; Neoadjuvant Therapy; Drug Resistance, Neoplasm; Hypoxia
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body; Esophageal Neoplasms; Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Hypoxia | interventions — pembrolizumab; Paclitaxel; Cisplatin

STUDY DESIGN:
Intervention Model Description: Pembrolizumab in combination with chemotherapy (Paclitaxel plus Cisplatin, TP regimen)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab + Chemo (Experimental): Neoadjuvant setting (Pembrolizumab in combination with chemotherapy): Up to 4 cycles concurrent administrations of (1) Paclitaxel, which are administrated intravenously at 150 mg/m^2 dosage on Day 1 of each 3-week cycle; (2) Cisplatin, which are administrated intravenously at 80 mg/m^2 dosage on Day 1 of each 3-week cycle; (3) Pembrolizumab, which are administrated intravenously at 200 mg dosage on Day 1 of each 3-week cycle.
  Adjuvant setting (Pembrolizumab in combination with chemotherapy): All participants who are assessed as ineligible or unnecessary for surgery after neoadjuvant treatment may be eligible for up to an additional 17 cycles (approximately 1 year) of Pembrolizumab treatment in combination with chemotherapy.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — Biological: Pembrolizumab 200 mg administered IV Q3W on Day 1 of each 3-week cycle, up to 4 administrations in neoadjuvant setting.
  Other Names: Keytruda; MK-3475
Drug: Paclitaxel — Drug: Paclitaxel 150 mg/m^2 administered IV Q3W on Day 1 of each 3-week cycle, up to 4 administrations in neoadjuvant setting.
Drug: Cisplatin — Drug: Cisplatin 80 mg/m^2 administered IV Q3W on Day 1 of each 3-week cycle, up to 4 administrations in neoadjuvant setting.

SUMMARY:
The purpose of this trial is to evaluate efficacy and safety of pembrolizumab plus standard of care (SOC) chemotherapy with cisplatin and paclitaxel as neoadjuvant treatment in participants with locally advanced esophageal squamous cell carcinoma (ESCC), and to explore treatment resistance mechanisms.

DETAILED DESCRIPTION:
The overall primary efficacy hypotheses are as follows:

In all eligible participants with locally advanced ESCC, pathologic complete response (pCR) rate is non-inferior with pembrolizumab plus SOC chemotherapy compared with historical benchmark.

The overall primary translational hypotheses are as follows:

Major hypoxia signals are significantly higher in baseline or post-treatment tumor samples from non-responders to pembrolizumab plus SOC chemotherapy, as compared to those samples from responders.

ELIGIBILITY:
Inclusion Criteria:

[Participants are eligible to be included in the study only if all of the following criteria apply]

1. Male/female participants who are at least 18 years of age on the day of providing documented informed consent with histologically or cytologically confirmed diagnosis of locally advanced and surgically resectable cT2-T4a NX M0 esophageal squamous cell carcinoma (ESCC) (per AJCC 8th edition) and who are previously untreated will be enrolled in this study.
2. Male participants:

   A male participant must agree to use a contraception during the treatment period and for at least 95 days after the last dose of study treatment and refrain from donating sperm during this period.
3. Female participants:

   A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
8. Have adequate organ function. Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

[Participants are excluded from the study if any of the following criteria apply]

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has had an allogenic tissue/solid organ transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate in all eligible participants with locally advanced ESCC | Up to approximately 6 months (1-September-2022 till 1-March-2023)
  Pathologic complete response is used as surrogate efficacy endpoint and is assessed by the Mandard tumor regression grade (TRG). PCR is defined as TRG1 plus no positive lymph node.
Major hypoxia signals in baseline or post-treatment tumor samples from all eligible participants with locally advanced ESCC | Up to approximately 12 months (1-September-2022 till 1-September-2023)
  Major hypoxia signals in tumor microenvironment (TME) are assessed by IHC methods, using tumor samples acquired pre- and post-treatment. Major hypoxia signals are to be compared between non-responders and responders to pembrolizumab plus SOC chemotherapy. In this neoadjuvant study, we define that patients who fail to reach major pathologic response (mPR) before surgery are classified as non-responders, and patients who reach mPR before surgery as responders. MPR is assessed by the Mandard TRG. MPR is defined as combined TRG1 and TRG2.

SECONDARY OUTCOMES:
PCR rate in eligible participants with locally advanced ESCC whose tumors are PD-L1 biomarker positive (CPS ≥1) | Up to approximately 12 months (1-September-2022 till 1-September-2023)
  Pathologic complete response is used as surrogate efficacy endpoint and is assessed by the Mandard tumor regression grade (TRG). PCR is defined as TRG1 plus no positive lymph node. PD-L1 expression is measured by 22C3 clone PD-L1 IHC assay followed by combined positive score (CPS) scoring methods.
Event-free survival (EFS) in the 3-year follow-up of all eligible participants with locally advanced ESCC | Up to approximately 48 months (1-September-2022 till 1-September-2026)
  EFS is defined as time from allocation to any of the following events: progression of disease that precludes surgery, local or distant recurrence, a second primary tumor, or death due to any cause.
Cell lineage-specific hypoxia signals in baseline or post-treatment tumor samples from all eligible participants with locally advanced ESCC | Up to approximately 12 months (1-September-2022 till 1-September-2023)
  Lineage-specific hypoxia signals in TME are assessed by multi-color flow cytometry in defined immune subsets and tumor, using surgical tumor samples acquired post-treatment. Lineage-specific hypoxia signals are to be compared between non-responders and responders to pembrolizumab plus SOC chemotherapy. In this neoadjuvant study, we define that patients who fail to reach mPR before surgery are classified as non-responders, and patients who reach mPR before surgery as responders. MPR is assessed by the Mandard TRG. MPR is defined as combined TRG1 and TRG2.

OTHER OUTCOMES:
Spatial proteomic measurement of hypoxia and defined cell lineages in baseline or post-treatment tumor samples from all eligible participants with locally advanced ESCC | Up to approximately 12 months (1-September-2022 till 1-September-2023)
  Spatial proteomic measurement of hypoxia and defined cell lineages are assessed by multiplex IHC assay.
Single cell genomic measurement of hypoxia pathway genes in post-treatment tumor samples from all eligible participants with locally advanced ESCC. | Up to approximately 12 months (1-September-2022 till 1-September-2023)
  Single cell genomic measurement of hypoxia pathway genes are assessed by single cell RNA sequencing.
PCR rate in eligible participants with locally advanced ESCC whose tumors are PD-L1 biomarker positive (CPS ≥10) | Up to approximately 12 months (1-September-2022 till 1-September-2023)
  PCR is used as surrogate efficacy endpoint and is assessed by the Mandard tumor regression grade (TRG). PCR is defined as TRG1 plus no positive lymph node. PD-L1 expression is measured by 22C3 clone PD-L1 IHC assay followed by CPS scoring methods.
R0 resection rate in all eligible participants with locally advanced ESCC | Up to approximately 12 months (1-September-2022 till 1-September-2023)
  R0 resection is defined as microscopically margin-negative resection, without remaining gross or microscopic tumor in the primary tumor bed.
EFS in eligible participants with locally advanced ESCC, stratified by PD-L1 biomarker expression (CPS ≥10, ≥1 and <1) | Up to approximately 48 months (1-September-2022 till 1-September-2026)
  EFS is defined as time from allocation to any of the following events: progression of disease that precludes surgery, local or distant recurrence, a second primary tumor, or death due to any cause. PD-L1 expression is measured by 22C3 clone PD-L1 IHC assay followed by CPS scoring methods.

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, M.D., Ph.D., Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Fudan University Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
Time Frame: Data will become available within three months after assay completion or request from MSD, and will be archived for 10 years.
Access Criteria: Requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
URL: http://engagezone.msd.com/ds_documentation.php